Dr. Khaled M. Aldahmani Endocrine Department, Tawam Hospital, Al-Ain, United Arab Emirates

February 17, 2021

Dear Authority,

Please find enclosed our manuscript entitled:

# Decline in Radioiodine use but not total thyroidectomy in thyroid cancer patients treated in United Arab Emirates- A Retrospective Study

In the United Arab Emirates (UAE), Thyroid Cancer represents the third most common malignancy in the population mostly occurring in the 3rd-4th decades of life and presenting as a localized disease. The management of Thyroid Cancer (TC) has significantly changed in the last decade with several guidelines around the world. These changes resulted in lower rates of total Thyroidectomy and Radioiodine administration in some parts of the world. But very little is known about the trend in Thyroid Cancer management in Middle East and North Africa (MENA) region.

In this study we aim to analyze the trends of TC characteristics and treatment modalities in patients presenting to the largest oncology center in the UAE over the last decade. In addition, we evaluate factors associated with the extent of surgery and RAI therapy.

We believe that this manuscript would be well-suited to be published as a case-controlled study. In submitting this manuscript for publication, we hope to highlight the evaluation of clinicopathological features and treatment modalities in Thyroid Cancer patients in the UAE. The significance of Nationality and Lymph Node Factor involvement in Surgery and RAI use. Most patients were diagnosed with localized Papillary Thyroid Cancer with no significant change in the extent of surgical approach but a substantial decline in RAI therapy administration over time.

We confirm that this manuscript has not been submitted elsewhere for publication. There was no financial support for this work and authors will cover publication fees when study is accepted for publication. All authors contributed to the writing of this manuscript, revised it critically for important intellectual content, and approve its submission. The authors have no actual or potential conflicts of interest to declare. Please address all correspondence concerning this manuscript to me at kmdahmani@seha.ae

Thank you for your consideration for this manuscript.

Sincerely,

Dr. Khaled M. Aldahmani

Endocrine Department,

Tawam Hospital,

Al-Ain, United Arab Emirates

kmdahmani@seha.ae

## Decline in Radioiodine use but not total thyroidectomy in thyroid cancer

## patients treated in United Arab Emirates- A Retrospective Study

## 3 Abstract

2

## 4 Background:

## 5 **Objectives:**

- 6 To assess the trend of clinicopathological features and treatment modalities in patients with
- 7 thyroid cancer (TC) in the largest oncology center in the United Arab Emirates (UAE).

## 8 **Methods:**

- 9 A retrospective analysis of patients with TC presenting to a tertiary care hospital in Al Ain,
- 10 UAE between September 2008 and December 2018 identified using ICD 9 & 10 codes was
- performed. Data on demographics, histopathology, surgical extent, and use of Radioiodine
- 12 (RAI) were extracted. Exact logistic and ordinal logistic regressions were performed to analyze
- the annual trend in features and management of TC, and logistic regression analysis was
- 14 performed to identify predictors of total thyroidectomy and RAI use.

#### 15 **Results:**

- A total of 762 patients were included in the analysis (mean age:  $39.6 \pm 12.6$  years, 45 (60%)
- women). The majority (92.2%) were diagnosed with papillary thyroid cancer (PTC) and 83.9%
- had tumor size of < 4 cm. All patients underwent surgery (93.8% total thyroidectomy, 6.2%
- lobectomy) and 77.4% received RAI therapy overall with a significant (p<0.001) decline from
- 20 100% in 2008 to 60% in 2018. In multivariate analysis, nationality, and lymph node (LN)
- 21 involvement were significant predictors of total thyroidectomy, while nationality, LNs, year of
- diagnosis, and tumor size significantly predicted RAI use.

## 23 Conclusion:

- 24 Most patients in our cohort were diagnosed with localized PTC with no significant change in
- 25 the extent of surgical approach but a substantial decline in RAI therapy administration over
- 26 time. Nationality and LN involvement were significant predictors of surgical extent and RAI
- 27 use.

## Introduction

28

29 Management of thyroid cancer (TC) has significantly changed in the last decade with several 30 guidelines advocating for a conservative approach in the majority of patients [1-2]. While these 31 changes resulted in lower rates of total thyroidectomy and radioiodine administration in some 32 parts of the world [3-4], data on TC from the Middle East and North Africa (MENA) region 33 has largely focused on incidence, characteristics, and treatment outcomes with recent 34 exploration of TC genetics [5-12]. Little is known about the trend in TC management in this 35 region. 36 It is difficult to predict if management of TC in the MENA region would follow similar trends 37 compared to other parts of the world. For example, it is unknown if patients or even physicians 38 are willing to observe micro papillary TC (MPTC) rather than offering surgery, at least 39 lobectomy. Similarly, attitudes toward the extent of surgery and use of RAI in localized TC 40 following the publication of the guidelines from the United Kingdom (UK) in 2014 and the 41 2015 American Thyroid Association (ATA) has not been well reported in the MENA region. 42 Furthermore, ethnicity has been shown to influence the incidence and outcomes of TC in some 43 studies [13-14]. Whether ethnicity impacts management of TC patients in our region remains 44 unclear. 45 In the United Arab Emirates (UAE), TC represents the third most common malignancy in the 46 population mostly occurring in the 3rd-4th decades of life and presenting as a localized disease 47 [15]. We aimed to study trends of TC characteristics and treatment modalities in patients 48 presenting to the largest oncology center in the UAE over the last decade. In addition, we 49 evaluated factors associated with the extent of surgery and RAI therapy.

50

51

53

54

55

56

57

58

59

#### **Materials and Methods**

## 52 Study setting

This study was conducted in Tawam hospital (TWM), which provides tertiary care services to patients in the UAE. It is the only center delivering radioactive iodine (RAI) therapy and radiotherapy in Al Ain city. Most TC patients are followed in designated TC clinics within the endocrinology division or less commonly through other clinics (surgery, radiation, or medical oncology). The hospital runs monthly multidisciplinary team-based discussions on patients with TC, wherein decisions regarding RAI treatment and dose selection are determined jointly by nuclear medicine physicians and endocrinologists.

## Study Design and participants

- 61 We retrospectively evaluated all patients with TC presenting to TWM during the period of 62 September 2008 and December 2018. The beginning of data collection (September 2008) 63 reflects the inception time of electronic medical records (EMRs) use in the hospital. Cases of 64 TC were extracted from the EMRs using the International Classification of Disease 9 & 10 65 codes (193 & c73). Other variables were demographic information, year of diagnosis, type of 66 TC, histopathological subtype, lymph node (LN) involvement, type of thyroid surgery, use of 67 RAI treatment, and radiation therapy. The extent of surgery, the exact details of histopathology, 68 and the RAI dose were retrieved from the respective specialty reports. Tumor staging was reported according to the 8<sup>th</sup> edition of the American joint committee on cancer (AJCC)/TNM 69
- 71 noninvasive follicular type PTC were excluded.

## 72 Ethical considerations

73 The study was approved by Al Ain Medical District Human Research Ethical Committee and

staging system [16]. Those with incorrect pathological diagnosis, incomplete data, or

74 consent was waved.

75

76

70

60

## STROCSS Compliance

77 This work has been reported in line with the STROCSS criteria [17].

## 78 Statistical Analysis

79 The data were extracted using Microsoft Excel 2015 and imported into Stata 16.0 for statistical 80 analysis. Continuous variables were described using means and standard deviations (±SD). Categorical variables were described as frequency distributions. Variables of clinical features 81 82 and management were cross tabulated with the year of diagnosis and exact logistic and ordinal 83 logistic regressions were performed to analyze the annual trend in features and management of 84 TC as appropriate. The results of relative trend were reported as odds ratio (OR) with an overall 85 p<sub>trend</sub>. The OR=1 indicated no change over years, OR <1 indicated a decline, while OR >1 86 indicated an increase over years. Simple and multiple logistic regression analysis were 87 performed to assess the unadjusted and adjusted association of management of TC (RAI, 88 surgical management) with age, gender, nationality, year of diagnosis, tumor subtype, and other 89 co-variates. The results of simple and multiple logistic regression were reported as odd ratios

(OR) and adjusted odds ratios (AOR) respectively with their corresponding 95% confidence intervals (CI) and p-values.

# 

## Results

## Overall patients' demographics

A total of 762 patients were included in the analysis (Table 1). The mean age at the diagnosis was 39.7 (±12.6) and 583 (76.5%) were women. The vast majority of patients (92.1%) were diagnosed with PTC. Of those, the histology subtype was available for 555 patients with the two most common being classical (73.5%) and invasive follicular variant (22.3%). About 83.8% of the patients (N=555) had a tumor size of <4cm at diagnosis. The stage of TC was documented in 590 patients. Of those, 523 (88.6%) patients were stage I while 23 (3.9%) were stage IV. All patients underwent surgery with the majority receiving (93.8%) total thyroidectomy and 566 (77.4%) RAI therapy.

Table 1: Characteristics of thyroid cancer patients (n=762)

| Demographics | N (%) / Mean (±SD) |
|---------------------------|--------------------|
| Age – years (n=762) | 39.7 (±12.6) |
| Gender (n=762) | |
| Female | 583 (76.5) |
| Male | 179 (23.5) |
| Nationality | |
| UAE | 349 (45.8) |
| Others | 413 (54.2) |
| Tumor size (n=551) | |
| ≤1 cm | 147 (26.7) |
| 1.1 - 1.9 cm | 188 (34.1) |
| $\geq 2 - 3.9 \text{ cm}$ | 127 (23.1) |
| ≥4 cm | 89 (16.1) |
| Tumor Type (n=762) | |
| PTC | 702 (92.1) |
| FTC | 35 (4.6) |
| MTC | 19 (2.5) |
| Anaplastic | 6 (0.8) |
| PTC Subtype (n=555) | |
| Classical | 408 (73.5) |
| Follicular | 124 (22.3) |
| Others | 23 (4.1) |
| Stage (n=590) | |
| I | 523 (88.6) |

| II | 35 (5.9) |
|--------------------------|------------|
| III | 9 (1.5) |
| IV | 23 (3.9) |
| Type of surgery (n=754) | |
| Hemithyroidectomy | 47 (6.2) |
| Total thyroidectomy | 707 (93.8) |
| RAI ablation (n= 731) | |
| Yes | 566 (77.4) |
| No | 165 (22.6) |
| Radiotherapy use (n=762) | 10 (1.3) |

MTC: Medullary Thyroid Cancer, FTC: Follicular Thyroid Cancer, PTC: Papillary Thyroid Cancer, RAI: Radioactive Iodine, UAE:

United Arab Emirates

N does not always make up to 762 due to missing data for some variables

## Thyroid cancer characteristics over 10 years

The annual number of TC patients substantially increased during the study period from 25 cases in 2008 to 106 cases in 2018. Compared to men, the increment was significantly higher in women (Fig. 1). PTC was the most common type with a gradual increase (p=0.674) from 88% in 2008 to 95% in 2018 (Table 2). Stage 1 Tumors represented the majority of TC patients in 2008 and also showed an insignificant (p=0.267) increase till 2018. During the study period, compared to non-PTC types, the proportion of patients with PTC increased by 11% on average (p=0.021). In contrast, patients presenting with advanced **TC** relatively decreased by 10% (p=0.022) compared to stage 1 cancer.

Figure 1: Incident cases of thyroid cancer between 2008 and 2018, overall and by gender



## Trend in surgery and RAI treatment

Total thyroidectomy showed a modest decline (p=0.409) from 100% in 2008 to 90.1% in 2018.

The RAI treatment showed a significant decline (<0.001) from 100.0% in 2008 to 60.4% in 2018 (Table 2).

Table 2: TC cases over years, overall and by characteristics

| | 2008 | 2009 | 2010 | 2011 | 2012 | 2013 | 2014 | 2015 | 2016 | 2017 | 2018 | OR<br>(Ptrend) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Overall | 25<br>(3.3) | 48<br>(6.3) | 36<br>(4.7) | 46<br>(6.0) | 80<br>(10.5) | 82<br>(10.8) | 83<br>(10.9) | 83<br>(10.9) | 82<br>(10.8) | 91<br>(11.9) | 106<br>(13.9) | |
| Gender | | | | | | | | | | | | |
| Female | 17<br>(68.0) | 37<br>(77.1) | 23<br>(63.9) | 39<br>(84.8) | 64<br>(80.0) | 61<br>(74.4) | 63<br>(75.9) | 67<br>(80.7) | 66<br>(80.5) | 65<br>(71.4) | 81<br>(76.4) | 0.99 |
| Male | 8<br>(32.0) | 11<br>(22.9) | 13<br>(36.1) | 7<br>(15.2) | 16<br>(20.0) | 21<br>(25.6) | 20<br>(24.1) | 16<br>(19.3) | 16<br>(19.5) | 26<br>(28.6) | 25<br>(23.6) | (0.777) |
| Nationality | | | | | | | | | | | | |
| UAE | 10<br>(40.0) | 16<br>(33.3) | 11<br>(30.6) | 23<br>(50.0) | 36<br>(45.0) | 43<br>(52.4) | 40<br>(48.2) | 44<br>(53.0) | 33<br>(40.2) | 43<br>(47.3) | 50<br>(47.2) | 0.96 |
| Others | 15<br>(60.0) | 32<br>(66.7) | 25<br>(69.4) | 23<br>(50.0) | 44<br>(55.0) | 39<br>(47.6) | 43<br>(51.8) | 39<br>(47.0) | 49<br>(59.8) | 48<br>(52.7) | 56<br>(52.8) | (0.155) |
| Stages | | | | | | | | | | | | |
| I | 6<br>(75.0) | 27<br>(81.8) | 24<br>(85.7) | 28<br>(80.0) | 40<br>(87.0) | 53<br>(88.3) | 57<br>(89.1) | 66<br>(91.7) | 72<br>(93.5) | 73<br>(89.0) | 77<br>(90.6) | 0.00 |
| II | (0.0) | 4<br>(12.1) | (10.7) | (2.9) | (6.5) | (5.0) | 4<br>(6.3) | 5 (6.9) | 4<br>(5.2) | 5 (6.1) | (3.5) | 0.90<br>(0.022) |
| III-IV | 2<br>(25.0) | 2<br>(6.1) | 1 (3.6) | 6<br>(17.1) | (6.5) | 4<br>(6.7) | 3 (4.6) | 1 (1.4) | 1 (1.3) | 4<br>(4.9) | 5 (5.9) | |
| | | | | | 6 | | | | | | | |

| Tumor size | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <1 cm | 3<br>(50.0) | 6<br>(20.7) | 2<br>(8.0) | 11<br>(32.3) | 13<br>(30.2) | 23<br>(41.8) | 22<br>(37.3) | 34<br>(49.3) | 29<br>(38.7) | 27<br>(34.6) | 20<br>(25.6) | |
| 1.1-1.9 cm | 1<br>(16.7) | 6<br>(20.7) | 10<br>(40.0) | 5<br>(14.7) | 6<br>(13.9) | 8<br>(14.5) | 8<br>(13.6) | 17<br>(24.6) | 13<br>(17.3) | 20<br>(25.6) | 20<br>(25.6) | 0.96 |
| 2.0-3.9 cm | 2<br>(33.3) | 11<br>(37.9) | 4<br>(16.0) | 15<br>(44.1) | 16<br>(37.2) | 15<br>(27.3) | 18<br>(30.5) | 11<br>(15.9) | 21<br>(28.0) | 19<br>(24.4) | 26<br>(33.3) | (0.142) |
| ≥4.0 cm | 0<br>(0.0) | 6<br>(20.7) | 9<br>(36.0) | 3<br>(8.8) | 8<br>(18.6) | 9<br>(16.4) | 11<br>(18.6) | 7<br>(10.1) | 12<br>(16.0) | 12<br>(15.4) | 12<br>(15.4) | |
| Tumor type | | | | | | | | | | | | |
| PTC | 22<br>(88.0) | 45<br>(93.7) | 32<br>(88.9) | 38<br>(82.6) | 70<br>(87.5) | 75<br>(91.5) | 78<br>(94.0) | 78<br>(94.0) | 79<br>(96.3) | 84<br>(92.3) | 101<br>(95.3) | 1.11 |
| Other | 3<br>(12.0) | 3<br>(6.3) | 4<br>(11.1) | 8<br>(17.4) | 10<br>(12.5) | 7<br>(8.5) | 5<br>(6.0) | 5<br>(6.0) | 3<br>(3.7) | 7<br>(7.7) | 5<br>(4.7) | (0.021) |
| PTC subtype | | | | | | | | | | | | |
| Classical | 13<br>(61.9) | 29<br>(69.1) | 28<br>(93.3) | 27<br>(77.1) | 54<br>(84.4) | 38<br>(62.3) | 40<br>(71.4) | 34<br>(66.7) | 43<br>(68.3) | 57<br>(80.3) | 45<br>(73.8) | 1.01 |
| Follicular | 7<br>(33.3) | 11<br>(26.2) | 2<br>(6.7) | 7<br>(20.0) | 8<br>(12.5) | 21<br>(34.4) | 13<br>(23.2) | 15<br>(29.4) | 16<br>(25.4) | 10<br>(14.1) | 14<br>(22.9) | (0.962) |
| RAI use | | | | | | | | | | | | |
| No | $0 \\ (0.0)$ | 2<br>(4.4) | 1<br>(2.78) | 6<br>(13.3) | 8<br>(10.1) | 12<br>(15.0) | 17<br>(21.5) | 22<br>(28.9) | 27<br>(34.6) | 30<br>(34.5) | 40<br>(39.6) | 0.75 |
| Yes | 25<br>(100.0) | 43<br>(95.6) | 35<br>(97.2) | 39<br>(86.7) | 71<br>(89.9) | 68<br>(85.0) | 62<br>(78.5) | 54<br>(71.1) | 51<br>(65.4) | 57<br>(65.5) | 61<br>(60.4) | (<0.001) |
| Surgical | | | | | | | | | | | | |
| management | | _ | _ | | _ | | | _ | _ | | | |
| Hemithyroidectomy | 0<br>(0.0) | (2.1) | 0<br>(0.0) | (0.0) | 2<br>(2.5) | 4<br>(4.9) | 6<br>(7.2) | 7<br>(8.4) | 3<br>(3.7) | (3.3) | 10<br>(9.5) | 0.89 |
| Thyroidectomy | 25<br>(100.0) | 47<br>(97.9) | 36<br>(100.0) | 46<br>(100.0) | 78<br>(97.5) | 78<br>(95.1) | 77<br>(92.8) | 76<br>(91.6) | 79<br>(96.3) | 88<br>(96.7) | 95<br>(90.5) | (0.054) |

OR: Odds Ratio, RAI: Radioactive Iodine

P-values are estimated for Exact logistic regression and ordinal logistic regression

Tumor size

## **Correlates of Surgery and RAI treatment**

In multiple logistic regression, non-UAE national patients were more likely to require total thyroidectomy (OR: 2.46 [CI: 1.21 - 4.94]). No other significant correlates of surgical extent were identified (Table 3).

Table 3. Simple and multiple logistic regression analysis of surgical management of thyroid cancer with selected variables.

| Variables | With Total<br>Thyroidectomy | Unadjusted A | nalysis | Adjusted Analysis | |
|---|---|---|---|---|---|
| | n (%) | OR (95% CI) | P-value | AOR (95% CI) | P-value |
| Year | | | | | |
| 2008-2010 | 107 (98.2) | Reference | | Reference | |
| 2011-2013 | 195 (93.7) | 0.28 (0.06 - 1.26) | 0.098 | 1.06 (0.10 - 10.93) | 0.962 |
| 2014-2016 | 230 (92.7) | 0.24 (0.05 - 1.05) | 0.058 | 0.33 (0.04 - 2.83) | 0.314 |

| 2017-2018 | 175 (92.6) | 0.23 (0.05 - 1.05) | 0.058 | 0.40 (0.05 - 3.48) | 0.407 |
|---|---|---|---|---|---|
| Age – Mean ±SD | $39.5 \pm 12.3$ | 0.99 (0.97 - 1.02) | 0.612 | 1.01 (0.97 - 1.05) | 0.653 |
| Sex | | | | | |
| Female | 542 (93.6) | Reference | | Reference | |
| Male | 165 (94.3) | 1.13 (0.55 - 2.31) | 0.746 | 0.60 (0.19 - 1.89) | 0.386 |
| Nationality | | | | | |
| UAE | 315 (90.5) | Reference | | Reference | |
| Others | 392 (96.5) | 2.93 (1.54 - 5.58) | 0.001 | 5.82 (1.85 - 18.30) | 0.003 |
| PTC Subtype | | | | | |
| Other | 22 (95.7) | Reference | | Reference | |
| Classical | 388 (95.6) | 0.98 (0.13 - 7.68) | 0.985 | 1.14 (0.13 - 10.45) | 0.907 |
| Follicular | 117 (94.3) | 0.76 (0.09 - 6.49) | 0.802 | 1.01 (0.10 - 9.88) | 0.992 |
| Tumour size | | | | | |
| ≤ 1.0 cm | 166 (88.8) | Reference | | Reference | |
| 1.1-1.9 cm | 111 (95.7) | 2.81 (1.03 - 7.66) | 0.044 | 2.05 (0.55 - 7.69) | 0.285 |
| 2.0-3.9 cm | 148 (94.3) | 2.08 (0.92 - 4.68) | 0.077 | 1.43 (0.45 - 4.51) | 0.540 |
| $\geq 4.0 \text{ cm}$ | 85 (95.5) | 2.69 (0.89 - 8.08) | 0.078 | 1.99 (0.45 - 8.75) | 0.362 |
| Lymph node | | | | | |
| No | 384 (91.4) | Reference | | Reference | |
| Yes | 156 (97.5) | 3.66 (1.28 - 10.44) | 0.015 | 2.74 (0.74 - 10.15) | 0.131 |

AOR: Adjusted Odds Ratio, CI: Confidence Interval, OR: Odds Ratio, PTC: Papillary Thyroid Cancer, RAI: Radioactive Iodine, SD: Standard Deviation, UAE: United Arab Emirates

Multiple logistic regression analysis showed that compared to 2008-2010, the likelihood of receiving RAI was 58% less in 2011-2013, 84% less in 2014-2016, and 92% less in 2017-2018. In addition, non-UAE nationals, those with larger tumor sizes, and LN involvement were more likely to receive RAI treatment (Table 4).

Table 4. Simple and multiple logistic regression analysis of RAI with selected covariates.

| 1 | 52 |
|---|----|
| 1 | 53 |

| Variables | With RAI | Unadjusted Aı | ıalysis | Adjusted An | alysis |
|---|---|---|---|---|---|
| | n (%) | OR (95% CI) | P-value | AOR (95% CI) | P-value |
| Year | | | | | |
| 2008-2010 | 103 (97.2) | Reference | | Reference | |
| 2011-2013 | 178 (87.3) | 0.20 (0.06 - 0.67) | 0.010 | 0.42 (0.11 - 1.52) | 0.187 |
| 2014-2016 | 167 (71.7) | 0.07 (0.10 - 0.24) | < 0.001 | 0.16 (0.05 - 0.54) | 0.003 |
| 2017-2018 | 118 (62.8) | 0.05 (0.02 - 0.16) | < 0.001 | 0.08 (0.02 - 0.29) | < 0.001 |
| Age – Mean ±SD | $39.5 \pm 12.6$ | 0.99 (0.98 - 1.01) | 0.172 | 0.99 (0.98 - 1.02) | 0.950 |
| Sex | | | | | |
| Female | 423 (75.8) | Reference | | Reference | |
| Male | 143 (82.7) | 1.52 (0.98 - 2.36) | 0.061 | 1.15 (0.64 - 2.05) | 0.650 |
| Nationality | | | | | |
| UAE National | 243 (73.2) | Reference | | Reference | |
| Other national | 323 (80.9) | 1.56 (1.10 - 2.21) | 0.013 | 1.63 (1.04 - 2.56) | 0.033 |
| Diagnosis | | | | | |

| Others | 39 (67.2) | Reference | | Reference | |
|---|---|---|---|---|---|
| PTC | 527 (78.3) | 1.76 (0.99 - 3.13) | 0.056 | 1.82 (0.62 - 5.38) | 0.276 |
| Tumour size | | | | | |
| $\leq 1.0$ cm | 99 (54.1) | Reference | | Reference | |
| 1.1-1.9 cm | 81 (73.0) | 2.29 (1.38 - 3.81) | 0.001 | 2.22 (1.26 - 3.89) | 0.005 |
| 2.0-3.9 cm | 130 (85.0) | 4.80 (2.82 - 8.15) | < 0.001 | 4.66 (2.59 - 8.41) | < 0.001 |
| ≥ 4.0 cm | 78 (92.9) | 11.03 (4.58 - 26.59) | < 0.001 | 9.82 (3.68 - 26.18) | < 0.001 |
| Stage | | | | | |
| I | 367 (72.7) | Reference | | Reference | |
| II | 30 (90.9) | 3.76 (1.13 - 12.52) | 0.031 | 0.77 (0.19 - 3.19) | 0.715 |
| III-IV | 22 (71.0) | 0.92 (0.41 - 2.04) | 0.836 | 0.58 (0.10 - 3.25) | 0.633 |
| Lymph node | | | | | |
| No | 280 (68.3) | Reference | | Reference | |
| Yes | 135 (87.7) | 3.30 (1.95 - 5.57) | < 0.001 | 3.55 (1.86 - 6.78) | < 0.001 |

AOR: Adjusted Odds Ratio, CI: Confidence Interval, OR: Odds Ratio, PTC: Papillary Thyroid Cancer, RAI: Radioactive Iodine, SD: Standard Deviation, UAE: United Arab Emirates

PTC represented the most common type of TC (92.1%) in our study with the majority having a

#### **Discussion**

154 155

156

157

158

159

160

161

162

163

164

165

166

167

168

169

170

171

172

173

174

175

176

classical subtype. Follicular TC was found in 4.6% of the patients while anaplastic and medullary cancers were rare. These findings are consistent with studies from the MENA region as well as other parts of the world [3-9]. The mean age at diagnosis of TC in our study was 39.7 years which is lower compared to the age of 44.7 years from a large retrospective study of 12, 508 TC patients diagnosed between 1972-2014 from 8 cancer registries in southeast china [18]. It is also lower that the mean age of 48 years from another retrospective study of 77, 276 TC patients diagnosed in the period of 1974-2013 using the surveillance, epidemiology and end results (SEER) cancer registry database in USA [19] or even from our same institution when 135 TC patients were studied between 1991-2005 [10]. However, the age at diagnosis was similar to data from a retrospective study of 600 TC patients diagnosed between 2004-2005 in nearby Saudi Arabia [7]. The proportion of patients with PTC subtype has increased during the study period, which is consistent with global data, although with a lower magnitude [19-20]. The proportion of advanced stage TC, however, decreased over the study period, which might be partly explained by the increased detection of localized TC cases. The later has been largely ascribed to the widespread use of imaging modalities to diagnose thyroid disorders and or other complaints from surrounding neck structures as well as the increased utilization of fine-needle aspiration to ascertain the nature of thyroid nodules [21-22]. This could also explain the increase in the annual number of TC evaluated in our centre. However, no conclusions can be drawn regarding

the temporal trend of TC, as our analysis was based on the absolute number of cases instead of rates.

The 2015 ATA guidelines suggest either lobectomy or total thyroidectomy for the management of TC for tumors 1-4 cm in size [2]. However, there is no universal consensus on the optimal surgical extent in TC management and significant variations are observed worldwide [23]. In our study, the majority of patients underwent total thyroidectomy (93.8%) with a small increase in hemi-thyroidectomy toward the last few years of the study. This finding is similar to another study retrospectively analyzing 44537 TC patients from SEER database between 2000-2014 in US and documenting a lower utilization of lobectomy in low-risk TC [24]. Of interest, cheng et al showed in 717 TC patients undergoing thyroidectomy between 2008-2016 that 44% of those initially eligible for lobectomy would need a completion surgery due to the presence of adverse histopathological features [25]. Similarly, kluijfohout *et al* evaluated 1000 patients with TC (size 1-4 cm) who underwent total thyroidectomy between 2000-2010 and reported that 122 out of 287 (43%) of patients who are eligible for lobectomy based on the 2015 ATA guidelines would need completion surgery due to the presence of high-risk features such as lymph node involvement (18%) and angioinvasion (12%) [26]. Therefore, determining the extent of surgery continues to be controversial with patient's preference and surgical expertise are paramount in the decision-making process. This issue is more apparent in microPTC, which represented about a quarter of our cohort where all patients underwent surgery. This is in variance with the growing evidence supporting active surveillance as a viable option in the majority of those patients [27-29].

Traditionally, RAI was administered to a large proportion of TC patients following total thyroidectomy. Subsequently, several but not all studies showed a limited benefit of RAI in low- to intermediate-risk groups in reducing disease-related recurrence and or mortality [30-31]. Therefore, the decline in the use of RAI has been advocated for by many TC management guidelines. Consistent with this, we noted a substantial decline in the use of RAI from 100% in 2008 to 60% in 2018. Similarly, Park *et al* showed a decline in RAI administration in 2015 compared to 1999 mostly in patients with localized disease [4]. Moreover, Sia *et al* reported a decline in RAI use from 76.6% in 2002-2006 to 26.8% in 2017-2018 mostly in low-risk patients [5]. The majority of our patients had tumor of <2cm in size with a limited number presenting with advanced disease (1.9% Stage IV), suggesting overuse of RAI. However, data on RAI indication in our study was not captured, therefore, precluding firm conclusions. Additionally,

209 variation in RAI use is well reported in many countries such as the US and Canada [32-33]. Of 210 interest, the use of RAI for example in T1 disease with unknown or negative lymph node status varied between 15 – 83% among different centers in Canada [33]. This wide variation in RAI 211 212 use underscores the limited data and uncertainty in the management of a significant proportion 213 of TC patients, necessitating the need for high-quality studies with long term follow up data to 214 confidently guide management in such patients. 215 The odds of undergoing total thyroidectomy and or receiving RAI ablation were higher in non-216 UAE nationals. This finding of ethnic variation in management of TC is intriguing and not well 217 reported in the literature. It might stem from the perceived risk of aggressive disease in certain 218 ethnicities. Lo et al retrospectively evaluated 723 patients with TC from Philippines with 5 219 years mean follow up and reported higher frequency of aggressive disease at presentation as 220 well as higher recurrence risk [34]. Furthermore, another study from the USA reported a higher 221 rate of adverse histology (microscopic extrathyroidal extension) in Chinese immigrants 222 compared to the non-Asian population [13]. Moreover, Tang et al retrospectively analyzed 223 70346 patients with TC from SEER database between 2004-2014 and showed worse overall 224 prognosis for black Americans with TC compared to white Americans [14]. Another factor 225 explaining this racial difference in the therapy might relate to the uncertainty in establishing 226 long-term follow-up plans in our country as 90% of the populations are non-nationals and many 227 of whom are workers with temporary living plans, which tempts the treating physician to adopt 228 an initial aggressive management strategy [35]. It would be interesting to explore which 229 ethnicity had advanced disease and or received aggressive therapy, but this information was not 230 captured in this study. Additional larger studies with long-term follow-up outcome data would 231 be important to clarify disease behaviour among different ethnicities.

Lymph node involvement in patients with TC is associated with increased recurrence risk and mortality [36]. Therefore, it is not surprising for lymph node involvement to be a predictor for RAI ablation as seen in our study. Tumour size was not associated with the extent of surgery in our study, perhaps due to the low number of patients undergoing lobectomy. However, it was associated with the need for RAI ablation. In 2015 ATA guidelines, tumor size is not an indication for RAI ablation in the absence of other adverse features [2]. Nonetheless, it is reassuring that the use of RAI has declined steadily during the study.

232

233

234

235

236

237

238

239

240

Our study has strengths and limitations. It is the first study in the MENA region to describe trends in TC characteristics and management patterns following publications of professional

TC management guidelines using a large number of patients. The main limitations of the study relate to its retrospective nature with incomplete documentation of data that could alter the decision of surgery and RAI such as the family history of TC, radiation exposure, and the number and size of involved lymph nodes. In addition, the reasons for determining the extent of surgery and the need/dose of RAI were not consistently recorded. Also, this study reflects the experience from a large referral center and may not be generalizable to other centers in the country.

## **Conclusion**

In summary, there is a substantial increase in the annual number of TC patients evaluated in our centre with the majority having PTC and stage 1 disease at diagnosis. Nationality and LN involvement were independent predictors of total thyroidectomy, while the year of diagnosis, nationality, LN involvement, and tumor size were predictors of RAI use. More studies are needed to understand factors affecting variation in TC management UAE.

255 Acknowledgement 256 The authors would like to thank Mr. Anvar Kandanath for data preparation and management. 257 258 **Disclosure Statement** 259 The authors have no conflicts of interest to declare. 260 261 **Funding Source** 262 There was no financial support for this work. 263 264 **Author Contributions** 265 M.A., A.S., A.M., E.A., A.K.M. conceived and wrote the manuscript. A.F. performed the 266 statistical analysis. A.F., S.R., A.O.H. revised the manuscript for important intellectual 267 content. All authors reviewed and approved the final manuscript. 268 269 270 Provenance and peer review 271 Not commissioned, externally peer-reviewed

## References

- 1. Perros P, Boelaert K, Colley S, Evans C, Evans RM, Gerrard Ba G, et al. Guidelines for the management of thyroid cancer. Clin Endocrinol (Oxf) 2014;81 Suppl 1:1–122.
- 2. Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, et al. American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016; 26(1):1–133. doi: 10.1089/thy.2015.0020.
- 3. Park KW, Wu JX, Du L, Leung AM, Yeh MW, Livhits MJ. Decreasing use of radioactive iodine for low-risk thyroid cancer in California, 1999 to 2015. J Clin Endocrinol Metab. 2018;103(3):1095–1101.
- 4. Sia Y, Dave RV, Nour D, Miller JA, Skandarajah AR, Tasevski R. Radioactive iodine ablation post differentiated thyroid cancer surgery: an analysis of use and impact of the American Thyroid Association guidelines. ANZ J Surg. 2019;89(11):E502-E506. doi:10.1111/ans.15522
- 5. Pambinezhuth F, Al Busaidi N, Al Musalhi H. Epidemiology of Thyroid Cancer in Oman. Ann Endocrinol Metab 2017; 1(1):11-17. doi: 10.36959/433/561.
- 6. Benouis A, Bekkouche Z, Merad, MS, Loudjedi L, Khelil H, Berber N. (2017) Thyroid Cancer in Western Algeria: Histopathological and Epidemiological Study. JCT 2017; 8:672-82. doi: 10.4236/jct.2017.87058.
- 7. Alzahrani AS, Alomar H, Alzahrani N. Thyroid cancer in Saudi Arabia: a histopathological and outcome study. Int J Endocrinol 2017; 1–7. doi: 10.1155/2017/8423147.
- 8. Safavi A, Azizi F, Rozita Jafari R, Chaibakhsh S, Safavi AA. Thyroid Cancer Epidemiology in Iran: a Time Trend Study. Asian Pac J Cancer Prev 2016;17(1):407-12. doi: 10.7314/apjcp.2016.17.1.407.
- 9. Ahmed RA, Aboelnaga EM. Thyroid cancer in Egypt: histopathological criteria, correlation with survival and oestrogen receptor protein expression. Pathol Oncol Res 2015; 21:793-802. doi: 10.1007/s12253-014-9892-5.
- 10. Al-Zaher N, Al-Salam S, El Teraifi H. Thyroid carcinoma in the United Arab Emirates: perspectives and experience of a tertiary care hospital. Hematol Oncol Stem Cell Ther 2008; 1(1):14–21. doi: 10.1016/S1658-3876(08)50055-0.
- 11. Al-Salam S, Sharma C, Afandi B, Al Dahmani K, Al-Zahrani AS, Al Shamsi A, et al. (2020) BRAF and KRAS mutations in papillary thyroid carcinoma in the United Arab Emirates. PLoS ONE 15(4): e0231341. https://doi.org/10.1371/journal.pone.0231341
- 12. Alzahrani AS, Alswailem M, Alswailem AA, Al-Hindi, Goljan E, Alsudairy N, et al. Genetic Alterations in Pediatric Thyroid Cancer Using a Comprehensive Childhood Cancer Gene Panel, J Clin Endocrinol Metab., dgaa389, https://doi.org/10.1210/clinem/dgaa389.
- 13. Shah BR, Griffiths R, Hall SF. Thyroid cancer incidence among Asian immigrants to Ontario Canada: A population-based cohort study. Cancer 2017; 123(17):3320-25. doi: 10.1002/cancr.30746.
- 14. Tang J, Kong D, Cui Q, Wang K, Zhang D, Liao X, et al. Racial disparities of differentiated thyroid carcinoma: clinical behaviour, treatments, and long-term outcomes. World J Surg Oncol 2018; 16(1):45. doi: 10.1186/s12957-018-1340-7.
- 15. Statistics and Research Center. Cancer Incidence in United Arab Emirates annual report of the UAE national cancer registry. Ministry of Health and Prevention-2015

- 16. Tuttle RM, Haugen B, Perrier ND. 2017a Updated American Joint Committee on cancer/tumor-node-metastasis staging system for differentiated and anaplastic thyroid cancer (eighth edition): what changed and why? Thyroid 27 751–756.
- 17. Agha RA, Borrelli MR, Vella-Baldacchino M, Thavayogan R and Orgill DP, for the STROCSS Group. The STROCSS Statement: Strengthening the Reporting of Cohort Studies in Surgery. International Journal of Surgery 2017: 46:198-202.
- 18. Du L, Wang Y, Sun X, Li H, Geng X, Ge M, et al. Thyroid cancer: trends in incidence, mortality and clinical-pathological patterns in Zhejiang Province, Southeast China. BMC Cancer 18, 291 (2018). <a href="https://doi.org/10.1186/s12885-018-4081-7">https://doi.org/10.1186/s12885-018-4081-7</a>
- 19. Lim H, Devesa SS, Sosa JA, Check D, Kitahara CM. Trends in Thyroid Cancer Incidence and Mortality in the United States, 1974-2013. JAMA. 2017;317(13):1338–1348.doi:10.1001/jama.2017.2719
- 20. Kilfoy BA, Zheng T, Holford TR, Han X, Ward MH, Sjodin A, et al. International patterns and trends in thyroid cancer incidence, 1973-2002. Cancer Causes Control 2009; 20(5):525–31. doi: 10.1007/s10552-008-9260-4.
- 21. Haymart MR, Banerjee M, Reyes-Gastelum D, Caoili E, Norton EC. Thyroid Ultrasound and the Increase in Diagnosis of Low-Risk Thyroid Cancer. J Clin Endocrinol Metab. 2019 Mar 1;104(3):785-792. doi: 10.1210/jc.2018-01933.
- 22. Franceschi S, Vaccarella S. Thyroid cancer: An epidemic of disease or an epidemic of diagnosis? Int J Cancer 2015; 136(11):2738–9. doi: 10.1002/ijc.29311.
- 23. Kovatch KJ, Hoban CW, Shuman AG. Thyroid cancer surgery guidelines in an Era of De-Escalation. Eur J Surg Oncol. 2018 March; 44 (3):297-306.
- 24. James BC, Timsina L, Graham R, Angelos P, Haggstrom DA. Changes in total thyroidectomy versus thyroid lobectomy for papillary thyroid cancer during the past 15 years. Surgery 2019; 166(1):41-7. doi: 10.1016/j.surg.2019.01.007.
- 25. Cheng SP, Chien MN, Wang TY, Lee JJ, Lee CC, Liu CL. Reconsideration of tumor size threshold for total thyroidectomy in differentiated thyroid cancer. Surgery 2018; 164(3):504-10. doi: 10.1016/j.surg.2018.04.019.
- 26. Kluijfhout WP, Pasternak JD, Lim J, Kwon JS, Vriens MR, Clark OH, et al. Frequency of High-Risk Characteristics Requiring Total Thyroidectomy for 1-4 cm Well-Differentiated Thyroid Cancer. Thyroid 2016; 26(6):820-24. doi: 10.1089/thy.2015.0495.
- 27. Ito Y, Miyauchi A, Inoue H, Fukushima M, Kihara M, Higashiyama T, et al. An observational trial for papillary thyroid microcarcinoma in Japanese patients. World J Surg 2010;34:28–35.
- 28. Kwon H, Oh HS, Kim M, Park S, Jeon MJ, Kim WG, et al. Active surveillance for patients with papillary thyroid microcarcinoma: a single center's experience in Korea. J Clin Endocrinol Metab 2017;102:1917–1925.
- 29. Tuttle RM, Fagin JA, Minkowitz G, Wong RJ, Roman B, Patel S, et al. Natural history and tumor volume kinetics of papillary thyroid cancers during active surveillance. JAMA Otolaryngol Head Neck Surg. 2017;143(10):1015–1020.
- 30. Lamartina L, Durante C, Filetti S, Cooper DS. Low-risk differentiated thyroid cancer and radioiodine remnant ablation: a systematic review of the literature. J Clin Endocrinol Metab. 2015 May;100(5):1748-61. doi: 10.1210/jc.2014-3882.

- 31. Kim SK, Woo JW, Lee JH, Park I, Choe J, Kim J, et al. Radioactive iodine ablation may not decrease the risk of recurrence in intermediate-risk papillary thyroid carcinoma. Endocr Relat Cancer 2016;23:367-76. 10.1530/ERC-15-0572
- 32. Haymart MR, Banerjee M, Stewart AK, Koenig RJ, Birkmeyer JD, Griggs JJ. Use of radioactive iodine for thyroid cancer. JAMA. 2011;306(7):721–728.
- 33. Rachinsky I, Rajaraman M, Leslie WD, Zahedi A, Jefford C, McGibbon A, et al. Regional Variation across Canadian Centers in Radioiodine Administration for Thyroid Remnant Ablation in Well-Differentiated Thyroid Cancer Diagnosed in 2000-2010. J Thyroid Res. 2016;2016:2867916.
- 34. Lo TEN, Uy AT, Maningat PDD. Well-Differentiated Thyroid Cancer: The Philippine General Hospital Experience: Endocrinol Metab 2016; 31(1):72-9. doi: 10.3803/EnM.2016.31.1.72.
- 35. Al-Shamsi H, Jaafar H, Tirmazy SH, Elkhoury M, Azribi F, Jelovac D et al. The State of Cancer Care in the United Arab Emirates in 2020: Challenges and Recommendations, A report by the United Arab Emirates Oncology Task Force. Gulf jo Onco 2020;32: 71-78.
- 36. Wang LY, Ganly I. Nodal metastases in thyroid cancer: prognostic implications and management. Future Oncol 2016; 12(7):981-94. doi: 10.2217/fon.16.10.